CLINICAL TRIAL: NCT02126527
Title: Phase I Study of Auranofin and Sirolimus in Adult Patients With Non-Small Cell Lung Cancer
Brief Title: Auranofin and Sirolimus in Treating Patients With Advanced Solid Tumors or Recurrent Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1213; NCI-2013-01180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-001054; P30CA015083 (NIH)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Auranofin; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (auranofin and sirolimus) (Experimental): Patients receive auranofin PO QD and sirolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: auranofin; Drug: sirolimus; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: auranofin — Given PO
  Other Names: Ridaura
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I clinical trial studies the side effects and best dose of auranofin and sirolimus when given together in treating patients with non-small cell lung cancer. Immunosuppressive therapy, such as auranofin and sirolimus, may be an effective treatment for non-small cell lung cancer. Sirolimus may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving auranofin and sirolimus may be an effective treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of auranofin plus sirolimus (Cohort I).

II. To determine the confirmed response rate of auranofin plus sirolimus (Cohort II).

SECONDARY OBJECTIVES:

I. To describe the adverse event and toxicity profiles associated with this treatment combination.

II. To evaluate response, time to progression, progression-free survival (PFS), overall survival (OS), and time to treatment failure in patients treated with this treatment combination.

TERTIARY OBJECTIVES:

I. To evaluate tumor biomarkers of protein kinase C (PKC) and mammalian target of rapamycin (mTOR) signaling activity as predictors of clinical outcome (i.e. response, PFS, OS) for patients receiving auranofin/sirolimus therapy.

II. To evaluate the use of surrogate biomarkers of PKC and mTOR inhibition in peripheral blood lymphocytes (PBLs) as predictors of clinical outcome (i.e. response, PFS, OS) for patients receiving auranofin/sirolimus therapy.

OUTLINE: This is a cohort I, dose-escalation study followed by a cohort II study.

Patients receive auranofin orally (PO) once daily (QD) and sirolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Cohort I (dose escalation) only: Histologic proof of an advanced, solid tumor that is now unresectable
* Cohort II (maximum tolerated dose) only:

  * Platinum-refractory non-small cell lung cancer (NSCLC) (platinum-refractory defined as either disease progression either during or within 6 months of completion of first-line platinum-based chemotherapy)
  * Measurable disease
* Evidence of disease progression =< 6 months prior to registration
* Received at least one prior approved chemotherapeutic regimen unless there is no known, approved therapeutic regimen for their malignancy
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets (PLT) >= 100,000/mm^3
* Total bilirubin =< 1.5 upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN (=< 5 x ULN for patients with liver involvement)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN (=< 5 x ULN for patients with liver involvement)
* Creatinine =< 1.5 x ULN
* Fasting blood glucose =< 126 mg/dL
* Fasting triglycerides =< 1.5 x ULN
* Fasting cholesterol =< 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to provide informed written consent
* Willing to return to Mayo Clinic in Florida for follow-up (during the active monitoring phase of the study); note: during the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Life expectancy >= 84 days (3 months)
* Willing to provide tissue and blood samples for correlative research purposes; note: the goals of this study include assessment of the biologic effects on surrogate markers of the agent(s) being tested and are, therefore, contingent upon availability of the biologic specimens
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 28 days prior to registration
  * Mitomycin C/nitrosoureas =< 42 days prior to registration
  * Immunotherapy =< 28 days prior to registration
  * Biologic therapy =< 28 days prior to registration
  * Radiation therapy =< 28 days prior to registration
  * Radiation to > 25% of bone marrow
  * Bevacizumab =< 28 days prior to registration
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV cardiovascular disease
* Central nervous system (CNS) metastases or seizure disorder; NOTE: patients with known brain metastases that have been successfully treated and stable for >= 6 months without requirement for corticosteroids and without seizure activity will be eligible
* Receiving therapeutic anticoagulation with warfarin; NOTE: prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices is allowed, provided that international normalized ratio (INR) < 1.5; therapeutic anti-coagulation with low molecular weight heparin is allowed at time of registration
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and/or patients known to be human immunodeficiency virus (HIV) positive
* Cohort II Only: Other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, patient must not be receiving other cytotoxic or molecularly targeted therapeutics treatment for their cancer; patients receiving certain hormonal manipulations as part of their treatment may be allowed to continue at the discretion of the principal investigator (PI) (e.g. luteinizing hormone-releasing hormone [LHRH] analogs for prostate cancer); concurrent endocrine therapy for breast cancer will not be permitted
* History of myocardial infarction or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias =< 168 days (6 months) prior to registration
* Known allergy to auranofin or other gold compounds
* Receiving any medications or substances that are strong inhibitors or strong inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); NOTE: use of strong inhibitors and inducers is prohibited =< 7 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
MTD defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Cohort I) | 28 days
Proportion of confirmed tumor responses assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Cohort II) | Up to 24 weeks
  Will be estimated by the number of confirmed responses divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Incidence of adverse events assessed using NCI CTCAE version 4.0 | Up to 2 years
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Overall toxicity incidence evaluated using the Common Toxicity Criteria (CTC) standard toxicity grading | Up to 2 years
  Overall toxicity incidence as well as toxicity profiles by dose level, patient, and tumor site will be explored and summarized. Frequency distributions, graphical techniques, and other descriptive measures will form the basis of these analyses.
Confirmed and best responses | Up to 2 years
  Will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall, by tumor group, and by cohort).
Time to progression | Up to 2 years
  Will be summarized descriptively using Kaplan Meier methodology, the log-rank test, and Cox Proportional Hazards models (where appropriate given the small sample size).
PFS | Up to 2 years
  Will be summarized descriptively using Kaplan Meier methodology, the log-rank test, and Cox Proportional Hazards models (where appropriate given the small sample size).
OS | Up to 2 years
  Will be summarized descriptively using Kaplan Meier methodology, the log-rank test, and Cox Proportional Hazards models (where appropriate given the small sample size).
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 2 years
  Will be summarized descriptively using Kaplan Meier methodology, the log-rank test, and Cox Proportional Hazards models (where appropriate given the small sample size).

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Menefee, M.D., Study Chair — Mayo Clinic campus in Florida
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States